CLINICAL TRIAL: NCT00156325
Title: A Double-Blind, Placebo-Controlled Trial of Escitalopram as a Mood Stabilizer for Bipolar II Disorder
Brief Title: Escitalopram as a Mood Stabilizer for Bipolar II Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 03283
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-01-02 (Estimated); Status verified 2005-09

CONDITIONS: Bipolar Disorders
Keywords: Bipolar Disorder; Depression; Hypomania; Mood Stabilizer
MeSH Terms: conditions — Bipolar Disorder; Depression; Mania | interventions — Escitalopram

INTERVENTIONS:
Drug: Escitalopram (Lexapro)

SUMMARY:
This study will investigate the efficacy of Escitalopram, a Selective Serotonin Reuptake Inhibitor (SSRI) antidepressant, in the treatment of Bipolar II Disorder.

The use of antidepressants for those with bipolar disorder appears common in clinical practice but is not countenanced - at least as monotherapy - in formal treatment guidelines. This view reflects concerns about the possibility of antidepressant drugs inducing switching and rapid cycling in those with Bipolar Disorder. Although the effectiveness of treating Bipolar II patients with SSRIs has received very little attention in the literature, observations of Bipolar II patients treated with SSRIs suggest they may have general mood stabilising properties. Many patients have reported improvements not only in their depressed mood, but also a reduction in the severity, duration and frequency of hypomanic episodes.

In this proof of concept study we specifically assess whether a standard dose of an SSRI antidepressant is more effective than placebo in reducing the frequency, severity and duration of both depressive and hypomanic episodes.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, cross-over trial of Escitalopram (10 mg) versus placebo (identical presentation) in subjects identified as having Bipolar II Disorder. The nine-month study will commence with a no-treatment baseline period of three months (Baseline Phase) to ensure that subjects meet criteria for episode frequency. Subjects compliant with and completing baseline period requirements will then be randomized to receive Escitalopram or placebo for three months (Phase 2) and will then subsequently cross over to receive the alternative compound for the final three-month period (Phase 3). Prior to that cross-over, there will be a two-day taper period to avoid potential withdrawal effects, followed by a seven-day wash-out period to avoid carry-over effects from drug to placebo. Subjects will be assessed at the start of the study, and every month thereafter for the entire nine-month period.

Subjects aged 18-65 meeting diagnostic criteria for Bipolar II disorder will be recruited. Diagnosis will be based on the Diagnostic and Statistical Manual of Mental Disorders with the exception of the minimum four-day duration criterion for hypomanic episodes. Subjects must have a minimum 2-year history of depressive and hypomanic episodes, with a mood disturbance (either 'high' or 'low') occurring at least monthly. Subjects will be excluded if they have previously been treated with anti-depressants or mood-stabilisers, or have a history of psychotic symptoms during episodes of either hypomania or depression. Subjects who are actively suicidal, have a significant personality disorder, substantive illicit drug use, or alcohol consumption >30g/day will also be excluded. Exclusion will also apply to subjects who are pregnant or breastfeeding, and those with a history of heart disease, liver disease, epilepsy or seizures.

Subjects will complete a number of self-report questionnaires about their mood and functioning on a monthly basis as well as monitoring their mood on a daily basis. A research psychologist or psychiatrist will complete (at monthly intervals) the Hamilton Depression Rating, Young Mania Rating Scale and the DSM-IV Social and Occupational Functioning Assessment Scale based on functioning over the previous week throughout the nine-month duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65
* Minimum two year history of depressive and hypomanic episodes
* Mood episodes occuring monthly
* Meet DSM-IV criteria for Bipolar II Disorder (with exception of minimum 4 day period for hypomanic episodes)

Exclusion Criteria:

* Previous treatment with any antidepressant, mood stabilizer or neuroleptic medication
* History of psychotic symptoms during hypomanic or depressive episodes
* Current suicidal behaviours
* Current substantive illicit drug use or alcohol consumption
* Significant personality disorder
* Pregnancy or breastfeeding
* History of heart disease, liver disease, epilepsy or seizures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2004-02; Study Completion 2005-02

PRIMARY OUTCOMES:
Frequency, Severity and duration of depressive and hypomanic episodes and impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Parker, Principal Investigator — Black Dog Institute/School of Psychiatry, University of New South Wales
Locations (1):
- University of New South Wales, Sydney, New South Wales, Australia